CLINICAL TRIAL: NCT05614063
Title: A Randomized, Double-blind, Placebo-Controlled, Multicenter Phase 3 Study to Evaluate the Safety, Tolerability, and Efficacy of XEN1101 as Adjunctive Therapy in Focal-Onset Seizures
Brief Title: A Randomized Study of XEN1101 Versus Placebo in Focal-Onset Seizures
Acronym: X-TOLE2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPF-010-301; 2022-502000-73-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Focal Onset Seizures
Keywords: Epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — XEN1101

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- XEN1101 25 mg/day (Experimental): XEN1101 25 mg/day
  Interventions: Drug: XEN1101
- XEN1101 15 mg/day (Experimental): XEN1101 15 mg/day
  Interventions: Drug: XEN1101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XEN1101 — XEN1101 Capsules
  Other Names: Azetukalner
  Arms: XEN1101 15 mg/day; XEN1101 25 mg/day
Drug: Placebo — Placebo Capsules
  Arms: Placebo

SUMMARY:
The X-TOLE2 Phase 3 clinical trial is a randomized, double-blind, placebo-controlled study that will evaluate the clinical efficacy, safety and tolerability of XEN1101 administered as adjunctive therapy in focal-onset seizures.

DETAILED DESCRIPTION:
Approximately 360 subjects will be randomized in a blinded manner to one of two active treatment groups or placebo in a 1:1:1 fashion (XEN1101 25 mg : 15 mg : Placebo). Eligible subjects will have up to 9.5 weeks of baseline to assess frequency of seizures, followed by 12 weeks of blinded treatment. In order to be included in the study, subjects must be treated with a stable dose of 1 to 3 allowable antiseizure medications (ASMs) for at least one month prior to screening, during baseline, and throughout the double-blind treatment period (DBP) of the study. During the DBP, subjects will be instructed to orally take XEN1101 or placebo once daily with an evening meal.

Subjects who complete the 12-week DBP will have the opportunity to qualify and enroll in a separate open-label extension (OLE) study for continued treatment with XEN1101. Subjects who do not enroll in the OLE will enter a 8-week post treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Be properly informed of the nature and risks of the study and give informed consent in writing, prior to entering the study
* Diagnosis (≥2 years) of focal epilepsy according to the International League Against Epilepsy (ILAE) Classification of Epilepsy (2017). Subject must have had adequate trials of at least 2 ASMs, which were given (and tolerated) at adequate therapeutic doses, without achieving sustained seizure freedom.
* Treatment with a stable dose of 1 to 3 allowable current ASMs for at least one month prior to screening, during baseline, and throughout the duration of the DBP
* Able to keep accurate seizure diaries

Exclusion Criteria:

* Previously documented electroencephalogram which shows any pattern not consistent with focal etiology of seizures.
* History of focal aware non-motor seizures only, non-epileptic psychogenic seizure, primary generalized seizure, developmental and epileptic encephalopathy, including Lennox-Gastaut syndrome.
* Seizures secondary to drug or alcohol use, ongoing infection, neoplasia, demyelinating disease, degenerative neurological disease, metabolic illness, progressive structural lesion, encephalopathy, or progressive central nervous system (CNS) disease.
* History of status epilepticus or repetitive seizures within the 12-month period preceding Visit 1 where the individual seizures cannot be counted.
* History of neurosurgery for seizures <1 year prior to Visit 1, or radiosurgery <2 years prior to enrollment.
* Any medical condition or personal circumstance that, in the opinion of the investigator, exposes the subject to unacceptable risk by participating in the study or prevents adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Median percent change (MPC) in monthly (28 days) focal seizure frequency from baseline to DBP for XEN1101 versus placebo. | From baseline through to the double blind period (week 12)

SECONDARY OUTCOMES:
Proportion of subjects experiencing ≥50% reduction in monthly (28 days) focal seizure frequency from baseline through the DBP for XEN1101 versus placebo. | From baseline through to the double blind period (week 12)
MPC in weekly (7 days) focal seizure frequency from baseline to Week 1 for XEN1101 versus placebo. | From baseline through to the week 1
Proportion of subjects experiencing "at least much improved" (including "much" and "very much improved") in Patient Global Impression of Change (PGI-C). | From baseline through to the double blind period (week 12)
To assess adverse events as criteria for safety and tolerability of XEN1101 | From screening through to 56 days post-final dose.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (127):
- United States (57):
  - Strada Patient Care Center, Mobile, Alabama
  - Xenoscience, Phoenix, Arizona
  - University of Arizona, Health Sciences Center, Tucson, Arizona
  - Clinical Trials, Inc, Little Rock, Arkansas
  - Brain Science Research Institute, Los Angeles, California
  - University of California, David Clinical & Translational Science Center Clinical Research (CCRC), Sacramento, California
  - Anschutz Health Sciences, Aurora, Colorado
  - Floridian Community Research Center, Coral Gables, Florida
  - Serenity Research, Miami, Florida
  - Research Institute of Orlando, LLC, Orlando, Florida
  - Panhandle Research & Medical Clinic, Pensacola, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Encore Medical Research of Weston, LLC, Weston, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy and Neurology, Boise, Idaho
  - Indiana University, IU Health Partners, Adult Neurology Clinic, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - University of Kentucky, Dept. of Neurology, Lexington, Kentucky
  - MaineHealth Neurology - Scarborough, Scarborough, Maine
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - MedStar Health Research Institute, Clinton, Maryland
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Cornwell Health, Grand Rapids, Michigan
  - Minneapolis Clinic of Neurology, Burnsville, Minnesota
  - Saint Louis University Medical School - Neurosciences Clinical Research Unit, St Louis, Missouri
  - Washington University, St. Louis, St Louis, Missouri
  - Northeast Epilepsy Group, Hackensack, New Jersey
  - Dent Neurosciences Research Center, Buffalo, New York
  - NYU Comprehensive Epilepsy Center (CEC), New York, New York
  - Weill Cornell Medicine/ New York-Presbyterian Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Onsite Clinical Solutions, LLC, Charlotte, North Carolina
  - Duke Neurology, Durham, North Carolina
  - Meridian Clinical Research, LLC, Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Providence Brain & Spine Institute, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Austin Epilepsy Care Center (AECC), Austin, Texas
  - ANESC Research, El Paso, Texas
  - UT Physicians Epilepsy Clinic, Houston, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Carilion Clinic - Neurology, Roanoke, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - University of Washington Main Hospital, Seattle, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (8):
  - INECO and Favoloro Fundation, Buenos Aires
  - Hospital General de Agudos J.M. Ramos Mejia, Buenos Aires
  - Hospital De Alta Complejidad en Red el Cruce Nestor Kirchner - SAMIC, Buenos Aires
  - STAT Research S.A., Buenos Aires
  - Hospital Italiano, Buenos Aires
  - CENyR, Caba
  - Hospital Córdoba, Córdoba
  - Sanatorio del Sur S.A., San Miguel de Tucumán
- Australia (9):
  - St Vincent's Hospital Melbourne, Fitzroy, Melbourne
  - The Royal Melbourne Hospital, Melbourne, Melbourne
  - Royal Prince Alfred Hospital (RAPH), Camperdown, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Southern Neurology, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The University of Queensland (UQ) - Mater Research Institute (MRI), Brisbane, Queensland
  - Austin Health Pharmacy Clinical Trials, Heidelberg, Victoria
  - The Alfred Hospital (Alfred Health), Melbourne, Victoria
- MHAT Puls AD, Blagoevgrad, Bulgaria
- Canada (3):
  - Center For Neurologic Research, Lethbridge, Alberta
  - London Health Sciences Centre, London, Ontario
  - Le Centre Hospitalier de l'Universite' de Montreal (CHUM), Montreal, Quebec
- Chile (2):
  - Centro de investigación Clinica UC, Santiago
  - Hospital Clínico Vina del Mar, Viña del Mar
- FORBELI s.r.o., Neurologicka ambulance, Prague, Czechia
- Georgia (2):
  - American Hospital Network LLC, Tbilisi
  - Institute of Neurology and Neuropsychology, Tbilisi
- Germany (8):
  - Epilepsy Center Bethel, Bielefeld
  - Universitatsklinikum Bonn, Bonn
  - Epilepsiezentrum Frankfurt Rhein-Main, Frankfurt
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Philipps-Universität Marburg, Marburg
  - LMU Munich, Department of Neurology, Munich
  - Universitätsklinikum Tübingen, Tübingen
  - Universitatsklinik fur neurologie, universitats - und Rehabilitationskliniken Ulm, Ulm
- Beaumont Hospital, Dublin, Ireland
- Italy (5):
  - Istituto delle Scienze Neurologiche di Bologna, Bologna
  - Università Degli Studi Gabriele d'Annunzio Di Chieti, Pescara
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Pediatrico Bambino Gesu, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome
- Latvia (2):
  - Pauls Stradina Clinical university hospital, Riga
  - Riga East University Hospital, Riga
- Mexico (2):
  - Human Science Research Trials S. de R.L. de C.V., Mexico City
  - Neurocencias Esudios Clinicos SC, Sinaloa
- New Zealand (2):
  - University of Auckland, Auckland
  - Waikato Hospital, Hamilton
- Poland (4):
  - Centrum Medyczne Neuromed, Bydgoszcz
  - NZOZ Novo-Med, Katowice
  - Twoja Przychodnia NCM, Nowa Sól
  - Neurosphera Sp. z o.o., Warsaw
- Portugal (3):
  - Unidade Local de Saúde de São João, Porto
  - Hospital Pedro Hispano, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, Santa Maria da Feira
- Spain (10):
  - Unitat d'Assaigs Clínics. Servei de Farmàcia, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Vithas La Milagrosa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - IIS-Fundacion Jimenez Diaz/Farmacia, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional De Malaga, Málaga
  - Hospital Universitario y Politecnico La Fe, Valencia
  - Hospital Clínico Universitario Valladolid, Valladolid
- United Kingdom (7):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospital of Wales, Cardiff
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - St. George's Hospital NHS Foundation Trust, London
  - Royal London Hospital for Integrated Medicine, London
  - John Radcliffe Hospital, Oxford
  - Northern Care Alliance NHS Foundation Trust, Salford Care Organisation, Salford

IPD SHARING:
Plan to Share IPD: No